CLINICAL TRIAL: NCT02019368
Title: A Randomized, Double-blind, Placebo Controlled, Crossover Study to Evaluate the Antioxidant Effect of Aged Garlic Extract in Heavy Smokers
Brief Title: Antioxidant Effect of Aged Garlic Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Wakunaga Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: eki-843
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Heavy Smoker or Non-smoker

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Smoker subjects take 6 capsules once a day for 4 weeks.
  Interventions: Dietary Supplement: Placebo
- Aged garlic extract (Experimental): Smoker subjects take 1.5 g of aged garlic extract in 6 capsules once a day for 4 weeks.
  Interventions: Dietary Supplement: Aged garlic extract
- Non-smoker (No Intervention): Oxidative status in non-smoker

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: Aged garlic extract
  Arms: Aged garlic extract

SUMMARY:
This is a randomized, double-blind, placebo controlled, crossover study to determine the antioxidant effect of aged garlic extract. This study will also compare the oxidative status in heavy smokers with that in non-smokers.

ELIGIBILITY:
Inclusion Criteria:

* Smoking (at least 20 cigarettes per day) or non-smoking (more than 20 years)

Exclusion Criteria:

* Under medication for chronic disease
* Garlic allergy
* Engaging in vigorous exercise
* Taking drugs or functional food that may possess antioxidant property
* Participation in any clinical trial within 90 days of the commencement of the trial
* Renal or hepatic dysfunction
* Heart disease

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Urinary 8-hydroxydeoxyguanosine (8-OHdG) | Every 4 weeks (Overall 12 weeks)

SECONDARY OUTCOMES:
High sensitive CRP | Every 4 weeks (Overall 12 weeks)
Blood pressure | Every 4 weeks (Overall 12 weeks)
Indices of the second derivative of photoplethysmogram (SDPTG) | Every 4 weeks (Overall 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Hiroshima, Japan